CLINICAL TRIAL: NCT00755703
Title: A Phase I, Dose-Ranging Safety and Immunogenicity Study of an Adenovirus-vectored Intranasal, Pandemic (Hemagglutinin H5) Influenza Vaccine, ADhVN1203/04.H5, in Healthy Adults
Brief Title: Safety and Immunogenicity Study of Adenovirus-vectored, Intranasal Pandemic Influenza Vaccine.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Altimmune, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Prevention
Other Study IDs: H-0701-2; #1-UCI-AI-06205-01
Record Dates: First submitted 2008-09-17; First posted 2008-09-19 (Estimated); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Influenza A Subtype H5N1 Infection
Keywords: Influenza; Vaccine; Pandemic; Avian influenza; Adenovirus strain 5; Vectored vaccine; Intranasal; Tissue-culture derived; Non-replicating
MeSH Terms: conditions — Influenza, Human; Influenza in Birds

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Group 1 (Experimental): There will be 12 subjects in Group 1 that will receive 10e8 viral particles of the Pandemic Influenza Vaccine administered via intranasal spray on day 0 and day 28 (+/- 4d).
  Interventions: Biological: Pandemic Influenza Vaccine
- Group 2 (Experimental): There will be 12 subjects in Group 2 that will receive 10e9 viral particles of the Pandemic Influenza Vaccine administered via intranasal spray on day 0 and day 28 (+/- 4d).
  Interventions: Biological: Pandemic Influenza Vaccine
- Group 3 (Experimental): There will be 12 subjects in Group 3 that will receive 10e10 viral particles of the Pandemic Influenza Vaccine administered via intranasal spray on day 0 and day 28 (+/- 4d).
  Interventions: Biological: Pandemic Influenza Vaccine
- Experimental: Group 4 (Placebo Comparator): There will be 12 subjects in Group 4 that will receive a placebo consisting of buffer administered via intranasal spray on day 0 and day 28 (+/- 4d).
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Pandemic Influenza Vaccine — Undetermined
  Arms: Group 1; Group 2; Group 3
Biological: Placebo
  Arms: Experimental: Group 4

SUMMARY:
The purpose of this study is to test the recombinant vaccine for safety and immunogenicity in healthy adults volunteers. Single dose, intranasally administered vaccine using an adenovirus-recombinant vector has provided a safe route for inducing protection in animals against pandemic influenza in preclinical studies.

The vaccine is non-replicating, tissue culture based and designed for intranasal delivery.

DETAILED DESCRIPTION:
Objectives:

The primary objective is to evaluate the safety of the AdhVN1203/04.H5 vaccine when administered intranasally in two doses with an interval of 28 days in healthy adults 19-49 years of age.

The secondary objective is to evaluated the immunogenicity of the AdhVN1203/04.H5 vaccine at three different doses (10e8, 10e9 and 10e10 viral particles) when administered intranasally in two doses with an interval of 28 days in healthy adults 19-49 years of age.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and females in good general health, 19-49 years of age
* Subjects must provide written consent
* Willing to participate through study completion
* Willing to undergo nasal washes and swabs and provide urine and blood samples per protocol for safety and immunogenicity analysis
* Female of child-bearing age must have a negative urine pregnancy test and be stable on a reliable means of contraception.
* Meet screening criteria for hematology, chemistry and urinalysis

Exclusion Criteria:

* Pregnant (or possibly pregnant) and lactating women
* Any flu/cold symptoms and/or fever greater than 101 degrees in 3 days prior to study enrollment
* Any intranasal steroid medication administered in the 10 days prior to study enrollment
* History of chronic rhinitis or presence of pre-existing nasal septal defects, nasal polyps or other gross abnormalities
* Any previous nasal cautery or significant surgery for nasal septal defects
* Any regular past or current use of intranasal illicit drugs or history of intravenous illicit drug use
* Asthma that is greater than mild in severity
* Diagnosed active Hepatitis B or C
* HIV positive at screening
* Known or suspected malignancy, leukemia, or lymphoma
* Immunosuppressed, altered or compromised immune status as a consequence of disease or treatment with systemic corticosteroids
* Receipt of an influenza vaccine within the past 6 months
* Receipt of any vaccine in the past 30 days
* Receipt of any investigational drug in the past 30 days
* Known Diabetes mellitus
* History of anaphylaxis or angioedema
* Hypertension that is not well controlled
* Any medical, psychiatric, or social condition, or occupational or other responsibility that, in the judgment of the investigator would serve to interfere or serve as a contraindication to, protocol adherence, assessment of safety or reactogenicity, or a participants's ability to give informed consent

Ages: 19 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2008-10; Primary Completion 2009-09 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
To assess the safety of a nasally administered adenovirus-vectored pandemic influenza vaccine in healthy human adults. | 56 day observations with 2 year follow-up

SECONDARY OUTCOMES:
Determination of immunogenicity and correlates of protection based on HI titers in vaccinates | 28 days and 56 days post vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Scott D. Parker, M.D., Principal Investigator — Alabama Vaccine Research Clinic, University of Alabama at Birmingham
Locations (1):
- Alabama Vaccine Research Center (UAB), Birmingham, Alabama, United States